CLINICAL TRIAL: NCT03203772
Title: Management of Pain in Limb Neuropathic Conditions Through Immersive Virtual Reality
Brief Title: Immersive Virtual Reality for Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5150437
Record Dates: First submitted 2017-06-05; First posted 2017-06-29 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Neuropathy; Phantom Limb Pain; Complex Regional Pain Syndromes; Neuropathic Pain
MeSH Terms: conditions — Phantom Limb; Complex Regional Pain Syndromes; Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Limb neuropathic conditions (Experimental): Includes phantom limb pain, complex regional pain syndrome
  Interventions: Other: Immersive Virtual Reality

INTERVENTIONS:
Other: Immersive Virtual Reality — Participants will engage in virtual visualization therapy in an immersive virtual reality environment

SUMMARY:
Investigating how neuropathic limb pain, including phantom limb pain or complex regional pain syndrome, is affected by virtual reality. While several studies have looked into virtual reality for treating this type of pain, few have used the latest immersive virtual reality hardware combined with motion control for an engaging virtual mirror therapy experience. The investigators are interested in studying the use of virtual reality as an alternative treatment option for these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of complex regional pain syndrome or phantom limb pain in an upper or lower limb

Exclusion Criteria:

* Cognitive impairment leading to inability to make own medical decisions
* Complete inability to utilize leg or arm muscles that are needed for motion controller tracking
* History of seizures within the last year

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-08-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of Virtual Reality Environment Use Questionnaire | Immediately following final virtual reality session
  Using a questionnaire, feedback over participant self-reported tolerance of the virtual reality environment, participant likelihood of recommending this therapy to others with similar conditions, reported sense of presence in presented scenario(s), comfort of virtual reality devices, impact on self-reported functional ability outside of clinic, and overall impression of virtual reality therapy will be recorded.
Pain Relief with Virtual Reality Therapy: Wong-Baker Scale | Change from initial scores prior to virtual reality exposure to immediately prior to and following virtual reality sessions, and up to 8 weeks following last sessions
  Change in Wong-Baker Faces pain scale will be measured. This will be done by obtaining pain scale scores immediately prior to therapy session, immediately following therapy, and several weeks post last therapy session.
Pain Relief with Virtual Reality Therapy: Visual Analog Scale | Change from initial scores prior to virtual reality exposure to immediately prior to and following virtual reality sessions, and up to 8 weeks following last sessions
  Change in Visual Analog Pain Scale will be measured. This will be done by obtaining pain scale scores immediately prior to therapy session, immediately following therapy, and several weeks post last therapy session.
Pain Relief with Virtual Reality Therapy: Short-Form McGill Pain Scale | Change from initial scores prior to virtual reality exposure to immediately prior to and following virtual reality sessions, and up to 8 weeks following last sessions
  Change in Short-Form McGill Pain Questionnaire will be measured. This will be done by obtaining pain scale scores immediately prior to therapy session, immediately following therapy, and several weeks post last therapy session.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chau, MD, Principal Investigator — Loma Linda Univeristy
Locations (1):
- Loma Linda University Health, East Campus Outpatient Rehabilitation Center, Loma Linda, California, United States